CLINICAL TRIAL: NCT03470688
Title: An Observational Study Designed to Investigate the Utilisation and Effectiveness of Originator and Biosimilar Anti-TNF Agents in Australian Rheumatology
Brief Title: Investigating the Utilisation and Effectiveness of Originator and Biosimilar Anti-TNF Agents
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Opal Rheumatology Ltd. (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: MSD biosimilars
Record Dates: First submitted 2018-03-06; First posted 2018-03-20 (Actual); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis; Ankylosing Spondylitis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Spondylitis, Ankylosing | interventions — MIDORI protein, mouse; Etanercept; Biosimilar Pharmaceuticals

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Originator: Originator anti-TNF agents. Dosage as per physician's decision based on approved indication.
  Interventions: Biological: Originator
- Biosimilar: Biosimilar anti-TNF agents. Dosage as per physician's decision based on approved indication.
  Interventions: Biological: Biosimilar

INTERVENTIONS:
Biological: Originator — Originator anti-TNF agents
  Other Names: Enbrel; All other originator anti-TNF agents
  Groups: Originator
Biological: Biosimilar — Biosimilar anti-TNF agents
  Other Names: Brenzys; All other anti-TNF biosimilars as they come to market
  Groups: Biosimilar

SUMMARY:
An observational study investigating the utilisation and effectiveness of originator and biosimilar anti-TNF agents in patients with rheumatoid arthritis, psoriatic arthritis, or ankylosing spondylitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of rheumatoid arthritis (RA), psoriatic arthritis (PsA) or ankylosing spondylitis (AS) who are being treated at a participating OPAL clinic.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female adults (>= 18 years) with a confirmed diagnosis of RA, PsA, or AS
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease activity score based on a 28 joint count (DAS28) | 3 years
  Comparative assessment of disease activity as measured by DAS28 in patients receiving originators vs biosimilars. Higher DAS28 scores indicate more severe disease activity.
Health Assessment Questionnaire Disability Index (HAQ-DI) | 3 years
  Comparative assessment of disease impact on quality of life and daily physical functions in patients receiving originators vs biosimilars. HAQ-DI is designed to measure impact on everyday life. Higher scores indicate more severe disability.

SECONDARY OUTCOMES:
36-item Short Form Health Survey (SF-36) | 3 years
  Comparative assessment of disease impact on quality of life in patients receiving originators vs biosimilars.
  The SF-36 uses 8 sub scales to assess patient vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health. Each sub scale is scored between 0-100, where lower scores indicate a greater impact on function.
Patient Health Questionnaire-2 (PHQ-2) | 3 years
  Comparative assessment of disease impact on the emotional health in patients receiving originators vs biosimilars, as measured by the PHQ-2.
  The PHQ-2 is a two-question survey to screen for depression, and higher scores indicate that the patient experienced depressed mood or anhedonia more frequently over the past two weeks.
Fatigue assessed by the Functional Assessment of Chronic Illness Therapy (FACIT) questionnaire | 3 years
  Comparative assessment of fatigue in patients receiving originators vs biosimilars, assessed using the FACIT-fatigue scale.
  FACIT-fatigue is a questionnaire used to measure fatigue levels in patients with rheumatoid arthritis. A higher score is associated with a greater level of fatigue.
Number of patients discontinuing the drug for safety reasons | 3 years
  Comparison between number of patients using originator vs biosimilar who discontinue therapy for safety reasons.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Bird, Principal Investigator — Optimus Research
Locations (22):
- Australia (22):
  - Canberra Rheumatology, Canberra, Australian Capital Territory
  - Rheumatology ACT, Canberra, Australian Capital Territory
  - Susan Street Specialists Centre, Camperdown, New South Wales
  - Hills Rheumatology, Castle Hill, New South Wales
  - Orthopaedic and Arthritis Centre, Chatswood, New South Wales
  - Georgetown Arthritis, Georgetown, New South Wales
  - Combined Rheumatology Practice, Kogarah, New South Wales
  - Rheumatology United, Penrith, New South Wales
  - Coast Joint Care, Maroochydore, Queensland
  - Gold Coast Rheumatology, Southport, Queensland
  - Townsville Hospital - Rheumatology, Townsville, Queensland
  - Hobart Specialists Group, Hobart, Tasmania
  - Rheumatology Tasmania, Hobart, Tasmania
  - Southern Rheumatology, Brighton, Victoria
  - Northern Rheumatology and Specialists, Brunswick, Victoria
  - Monash Rheumatology, Clayton, Victoria
  - Coburg Rheumatology, Coburg, Victoria
  - Melbourne Arthritis Associates, Fitzroy, Victoria
  - Footscray Specialist Rooms, Footscray, Victoria
  - Barwon Rheumatology Service, Geelong, Victoria
  - Peninsula Rheumatology, Langwarrin, Victoria
  - Subiaco Rheumatology, Subiaco, Western Australia